CLINICAL TRIAL: NCT03343301
Title: FIGHT: A Phase 3 Randomized, Double-Blind, Controlled Study Evaluating FPA144 and Modified FOLFOX6 in Patients With Previously Untreated Advanced Gastric and Gastroesophageal Cancer: Phase 2 Preceded by Dose Finding in Phase 1
Brief Title: A Study of Bemarituzumab (FPA144) Combined With Modified FOLFOX6 in Gastric/Gastroesophageal Cancer
Acronym: FIGHT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPA144-004 Phase 1
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Cancer; Gastrointestinal Cancer Metastatic; Gastric Cancer
Keywords: gastrointestinal cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bemarituzumab 6 mg/kg + mFOLFOX6 (Experimental): Participants received 6 mg/kg bemarituzumab administered every 2 weeks (Q2W) and mFOLFOX6 chemotherapy administered Q2W until unacceptable toxicity, disease progression, or death.
  Interventions: Biological: Bemarituzumab; Drug: Modified FOLFOX6
- Bemarituzumab 15 mg/kg + mFOLFOX6 (Experimental): Participants received 15 mg/kg bemarituzumab administered Q2W with a single additional bemarituzumab 7.5 mg/kg dose on cycle 1 day 8. Participants also received mFOLFOX6 chemotherapy administered Q2W. Treatment continued until unacceptable toxicity, disease progression, or death.
  Interventions: Biological: Bemarituzumab; Drug: Modified FOLFOX6

INTERVENTIONS:
Biological: Bemarituzumab — Administered by intravenous infusion over approximately 30 minutes
  Other Names: FPA144
Drug: Modified FOLFOX6 — Modified FOLFOX6 regimen consists of the following:
  * Oxaliplatin 85 mg/m² IV infusion over 120 minutes
  * Leucovorin 400 mg/m² IV infusion over 120 minutes, or 200 mg/m² levo-leucovorin if leucovorin is unavailable
  * 5-fluorouracil (5-FU) 400 mg/m² bolus over approximately 5 minutes then 5-FU 2400 mg/m² as a continuous IV infusion over approximately 48 hours.
  Other Names: mFOLFOX6

SUMMARY:
The primary objective of the phase 1 portion of this study is to determine the recommended dose of bemarituzumab in combination with 5-fluorouracil, leucovorin and oxaliplatin (modified FOLFOX6) to use in the phase 2 portion of the trial.

DETAILED DESCRIPTION:
Phase 1 is an open-label dose-escalation of bemarituzumab in combination with modified FOLFOX6 (mFOLFOX6). Eligible patients will have unresectable locally advanced or metastatic GI cancer of any type and be candidates to receive at least 2 doses of mFOLFOX6 chemotherapy. Phase 1 consists of 2 dosing cohorts of bemarituzumab in combination with mFOLFOX6 to determine the recommended dose of bemarituzumab in combination with mFOLFOX6 for the phase 2 portion of the study (see study record NCT03694522).

ELIGIBILITY:
Inclusion Criteria:

1. Disease that is unresectable, locally advanced, or metastatic (not amendable to curative therapy)
2. Understand and sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form (ICF) prior to any study-specific evaluation
3. Life expectancy of at least 3 months in the opinion of the investigator
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
5. Age ≥ 18 years at the time the ICF is signed
6. In sexually active patients (women of childbearing potential and males), willingness to use 2 effective methods of contraception, of which 1 must be a physical barrier method (condom, diaphragm, or cervical/vault cap) until 6 months after the last dose of FPA144. Other effective forms of contraception include:

   * Permanent sterilization (hysterectomy and/or bilateral oophorectomy, or bilateral tubal ligation with surgery, or vasectomy) at least 6 months prior to Screening
   * Women of childbearing potential who are on stable oral contraceptive therapy or intrauterine or implant device for at least 90 days prior to the study, or abstain from sexual intercourse as a way of living
7. Adequate hematological and biological function, confirmed by the following laboratory values within 96 hours prior to enrollment:

   Bone Marrow Function
   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Platelets ≥ 100 × 10^9/L
   * Hemoglobin ≥ 9 g/dL

   Hepatic Function
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 × upper limit of normal (ULN); if liver metastases, then < 5 × ULN
   * Bilirubin < 1.5 × ULN except in patients with Gilbert's disease

   Renal Function
   * Calculated creatinine clearance using cockcroft Gault formula ≥ 50 mL/min or estimated glomerular filtrate rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula ≥ 50 mL/min
8. International normalized ratio (INR) or prothrombin time (PT) < 1.5 x the ULN except for patients receiving anticoagulation, who must be on a stable dose of warfarin for 6 weeks prior to enrollment
9. Measurable or non-measurable, but evaluable disease using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
10. Histologically or cytologically confirmed GI malignancy for which mFOLFOX6 is considered an appropriate treatment (e.g., gastric cancer [GC], colorectal carcinoma, pancreatic adenocarcinoma)
11. Patient must be a candidate to receive at least 2 doses of mFOLFOX6 chemotherapy

Exclusion Criteria:

1. Untreated or symptomatic central nervous system (CNS) metastases (CNS imaging not required). Patients with asymptomatic CNS metastases are eligible provided they have been clinically stable for at least 4 weeks and do not require intervention such as surgery, radiation, or any corticosteroid therapy for management of symptoms related to CNS disease
2. Impaired cardiac function or clinically significant cardiac disease, including any of the following (Criteria a through g):

   1. Unstable angina pectoris ≤ 6 months prior to enrollment
   2. Acute myocardial infarction ≤ 6 months prior to enrollment
   3. New York Heart Association Class II-IV congestive heart failure
   4. Uncontrolled hypertension (as defined as ≥ 160/90 despite optimal medical management)
   5. Uncontrolled cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
   6. Active coronary artery disease
   7. Fridericia's corrected QT interval (QTcF) ≥ 480
3. Peripheral sensory neuropathy ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
4. Active infection requiring systemic treatment or any uncontrolled infection ≤ 14 days prior to enrollment
5. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known active or chronic hepatitis B or C infection
6. History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis)
7. Evidence or history of bleeding diathesis or coagulopathy
8. Radiotherapy ≤ 28 days of enrollment. Patients must be recovered from all acute radiotherapy-related toxicities. No radiopharmaceuticals (strontium, samarium) within 8 weeks of enrollment
9. Prior treatment with any selective inhibitor (e.g., AZD4547, BGJ398, JNJ-42756493, BAY1179470) of the fibroblast growth factor (FGF)-FGFR pathway
10. Ongoing adverse effects from prior systemic treatment > CTCAE Grade 1 (with the exception of Grade 2 alopecia)
11. Participation in another therapeutic clinical study or receiving any investigational agent within 28 days of enrollment or during this clinical study
12. Corneal defects, corneal ulcerations, keratitis, keratoconus, history of corneal transplant, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
13. Known positivity for human epidermal growth factor receptor 2 (HER2) (as defined by a positive immunohistochemistry [IHC] test of 3+ or IHC of 2+ with fluorescent in situ hybridization [FISH])
14. Major surgical procedures not permitted ≤ 28 days prior to enrollment. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before enrollment. In all cases the patient must be sufficiently recovered and stable before treatment administration
15. Women who are pregnant or breastfeeding (unless the patient is willing to interrupt breastfeeding during study treatment administration and then resume 6 months after study discontinuation); women of childbearing potential must not consider getting pregnant during the study
16. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, psychiatric disturbance, uncontrolled intercurrent illness including arterial thrombosis, or symptomatic pulmonary embolism)
17. Presence of any other condition that may increase the risk associated with study participation, or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry in the study
18. Known allergy, hypersensitivity or contraindication to components of the FPA144 formulation including polysorbate or to platinum-containing medications, 5-FU, or leucovorin
19. History of prior malignancy, except (Criteria a through f):

    1. Curatively treated non-melanoma skin malignancy
    2. Cervical cancer in situ
    3. Curatively treated Stage I uterine cancer
    4. Curatively treated ductal or lobular breast carcinoma in situ and not currently receiving any systemic therapy
    5. Localized prostate cancer that has been treated surgically with curative intent and presumed cured
    6. Solid tumor treated curatively more than 5 years previously without evidence of recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Marin Cancer Care, Greenbrae, California
  - Innovative Clinical Research Institute, Whittier, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Wilmont Cancer Institute, Rochester, New York
  - Tennessee Cancer Specialists, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study FPA144-004 was a Phase 1/2 study. Phase 1 was a safety run-in to determine the recommended dose of bemarituzumab to be administered in combination with a fixed dose of modified FOLFOX 6 (mFOLFOX6) chemotherapy regimen in the phase 2 part of the study. Phase 1 study results are reported herein; Phase 2 study details and results are reported separately (NCT03694522).
Pre-assignment Details: In Phase 1, dose cohorts were planned to begin at a bemarituzumab dose level of 6 mg/kg per dose, with enrollment into subsequent dose cohorts depending on safety and tolerability.
Groups:
- Bemarituzumab 6 mg/kg + mFOLFOX6: Participants received 6 mg/kg bemarituzumab administered every 2 weeks (Q2W) and modified FOLFOX6 (mFOLFOX6) chemotherapy administered Q2W until unacceptable toxicity, disease progression, or death.
Period: Overall Study
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Started | 3 | 9
Received Any Study Treatment | 3 | 9
Completed | 0 | 0
Not Completed | 3 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 2
Not completed — Other | 0 | 6
Not completed — Missing | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bemarituzumab 6 mg/kg + mFOLFOX6: Participants received 6 mg/kg bemarituzumab administered Q2W and mFOLFOX6 chemotherapy administered Q2W until unacceptable toxicity, disease progression, or death.
- Total: Total of all reporting groups
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6 | Total
Number analyzed (Participants) | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (21.46) | 62.3 (16.45) | 62.9 (16.78)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 1 | 5 | 6
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 9 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  White | 2 | 7 | 9
  Other | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status.
  * 0 = Fully active, able to carry out all pre-disease performance without restriction;
  * 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  * 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * 4 = Completely disabled, confined to bed or chair;
  * 5 = Dead.
  Participants
    0 (Fully active) | 0 | 6 | 6
    1 (Restricted activity but ambulatory) | 3 | 3 | 6
Anti-Cancer Treatment Prior to Enrollment [Count of Participants; unit: Participants]
  Yes | 2 | 7 | 9
  No | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events ≥ Grade 2
Description: A treatment-related adverse event (TRAE) is defined as an adverse event (AE) with an onset date on or after the date of first dose of study treatment, or an event present before treatment that worsened after treatment, and with an onset date prior to 28 days after the last date of dose, for which the investigator assessed as related to investigational product The investigator classified the severity of each AE using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0 on a scale from mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4), or death due to the AE (Grade 5).
Time Frame: From first dose of study drug up to 28 days after last dose; Actual median (min, max) duration of treatment emergent period was 19.3 (12.3, 22.3) weeks in the bemarituzumab 6 mg/kg group and 19.4 (4.0, 35.4) weeks in the bemarituzumab 15 mg/kg group.
Population: All participants who received any portion of at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 9
Participants | 1 | 4

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as any of the following events considered by the investigator to be related to study drug:
  * Absolute neutrophil count (ANC) < 0.5 × 10⁹/L > 5 days duration or febrile neutropenia.
  * Platelets < 25 × 10⁹/L or < 50 × 10⁹/L with bleeding requiring medical intervention or for > 3 days.
  * Grade 4 anemia.
  * Any Grade 2-3 ophthalmologic AE not resolving within 7 days.
  * Any Grade 4 ophthalmologic AE.
  * Any Grade 4 laboratory value.
  * Any Grade 3 laboratory values that are not of clinical significance according to investigator and Sponsor agreement if they do not resolve within 72 hours.
  * Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≥ 3× upper limit of normal (ULN) and concurrent total bilirubin ≥ 2× ULN not related to liver involvement with cancer.
  * Any non-hematological AE ≥ Grade 3 (except nausea, vomiting, and diarrhea).
  * Grade 3 nausea, vomiting or diarrhea not resolving with supportive care in 72 hours.
  * Grade 4 nausea, vomiting or diarrhea.
Time Frame: 28 days
Population: DLT-evaluable population includes all participants enrolled in Phase 1 of the study who received at least 2 doses of bemarituzumab (except for Cohort 2 [must have received 3 doses of bemarituzumab]) and mFOLFOX6 and completed Cycles 1 and 2 of treatment, or who experienced a DLT in Cycle 1 or Cycle 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 8
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events are defined as adverse events (AEs) that started or worsened between the start of study drug and 28 days after permanent discontinuation of study drug.
  A serious AE is defined as any untoward medical occurrence that at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability or incapacity;
  * Was a congenital anomaly or birth defect.
  The investigator assessed the causality/relationship between the study treatment and each AE, and assessed the severity of each AE according to the guidelines provided in NCI-CTCAE, version 5.0 on a scale from mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4), or death due to the AE (Grade 5).
  Ocular events associated with symptomatic corneal involvement and symptomatic and asymptomatic retinal involvement were events of special interest in this study.
Time Frame: From first dose of study drug up to 28 days after last dose; Actual median (min, max) duration of the treatment emergent period was 19.3 (12.3, 22.3) weeks in the bemarituzumab 6 mg/kg group and 19.4 (4.0, 35.4) weeks in the bemarituzumab 15 mg/kg group.
Population: All participants who received any portion of at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 9
Participants
  Any treatment-emergent adverse event (TEAE) | 3 | 9
  TEAE with Grade ≥ 3 | 1 | 6
  TEAE related to any study drug | 3 | 9
  TEAE related to bemarituzumab | 2 | 5
  TEAE related to any agent of mFOLFOX6 | 3 | 9
  TEAE with Grade ≥ 3 related to any study drug | 1 | 4
  Serious adverse event (SAE) | 0 | 4
  SAE related to any study drug | 0 | 1
  SAE related to bemarituzumab | 0 | 0
  SAE related to any agent of mFOLFOX6 | 0 | 1
  TEAE of special interest: corneal/retina | 0 | 4
  TEAE of special interest: corneal/retina related to bemarituzumab | 0 | 4
  TEAE of special interest: corneal/retina leading to discontinuation of bemarituzumab | 0 | 2
  TEAE leading to discontinuation of bemarituzumab | 0 | 4
  TEAE leading to discontinuation of any agent of mFOLFOX6 | 0 | 4
  TEAE leading to dose reduction of bemarituzumab | 1 | 0
  TEAE leading to dose reduction of any agent of mFOLFOX6 | 1 | 5
  TEAE leading to death (Grade 5) | 0 | 0

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Bemarituzumab
Time Frame: Cycle 1 day 1 at predose, 0.25, 4, 48, and 168 hours after end of infusion, and for participants in Cohort 2 day 8 at 0.25 and 4 hours end of infusion; Cycle 2 day 1 at predose, 0.25 and 48 hours after end of infusion.
Population: Participants who received bemarituzumab with available Cmax data
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 8
µg/mL
  Cycle 1 | 119 (8.52) | 329 (60.3)
  Cycle 2: number analyzed (Participants) | 3 | 7
  Cycle 2 | 123 (13.8) | 377 (82.8)

5. Secondary Outcome: Observed Serum Concentration of Bemarituzumab at the End of the Dose Interval (Ctrough)
Time Frame: Cycle 1 day 14 predose for cohort 1 and day 8 predose for cohort 2; Cycle 2 day 14 predose
Population: Participants who received bemarituzumab with available Ctrough data
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 8
µg/mL
  Cycle 1 | 16.5 (8.80) | 118 (25.1)
  Cycle 2 | 25.6 (10.6) | 131 (55.3)

6. Secondary Outcome: Area Under the Observed Concentration-time Curve From the Time of Dosing to Day 14 (AUC0-14)
Description: Area under the observed concentration-time curve from the time of dosing to Day 14 (0-336h) calculated by log-linear trapezoidal approximation.
Time Frame: Cycle 1 day 1 at predose, 0.25, 4, 48, and 168 hours after end of infusion, and for participants in Cohort 2 day 8 at 0.25 and 4 hours after the end of infusion.
Population: Participants who received bemarituzumab with available AUC data
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 7
μg*day/mL | 556 (232) | 2350 (394)

7. Secondary Outcome: Terminal Half-life (t1/2) of Bemarituzumab
Time Frame: Cycle 1 day 1 at predose, 0.25, 4, 48, and 168 hours after end of infusion, and for participants in Cohort 2 day 8 at 0.25 and 4 hours after end of infusion.
Population: Participants who received bemarituzumab with available half-life data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 3
days | 8.35 (3.36) | 4.23 (0.447)

8. Secondary Outcome: Number of Participants With Treatment Induced Anti-bemarituzumab Antibodies
Description: Postbaseline treatment induced antidrug antibody (ADA) positive is defined as participants with
  * ADA negative at baseline and ADA positive at any postbaseline timepoint, or
  * ADA positive at baseline and ADA positive with titer of at least 4-fold of the baseline titer at one or more postbaseline timepoint.
Time Frame: Samples were collected for ADA analysis predose on day 1 of Cycles 1, 2, 3, 7, and 10 and at 28 days following the last dose.
Population: The ADA-evaluable analysis set includes all enrolled participants who received at least 1 dose of bemarituzumab and had at least 1 ADA sample drawn at any timepoint with available ADA data.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
Number analyzed (Participants) | 3 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From enrollment to end of study; median (min, max) time on study was 19.4 (13.9, 22.4) weeks in Bemarituzumab 6 mg/kg + mFOLFOX6 and 28.6 (4.3, 49.6) weeks in Bemarituzumab 15 mg/kg + mFOLFOX6 group. Adverse Events: From first dose of any study drug to 28 days after last dose; Actual median (min, max) duration of treatment emergent period was 19.3 (12.3, 22.3) weeks in Bemarituzumab 6 mg/kg + mFOLFOX6 and 19.4 (4.0, 35.4) weeks in Bemarituzumab 15 mg/kg + mFOLFOX6 group.
Arm/Group | Bemarituzumab 6 mg/kg + mFOLFOX6 | Bemarituzumab 15 mg/kg + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/9
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemarituzumab 6 mg/kg + mFOLFOX6 (N=3) | Bemarituzumab 15 mg/kg + mFOLFOX6 (N=9)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bemarituzumab 6 mg/kg + mFOLFOX6 (N=3) | Bemarituzumab 15 mg/kg + mFOLFOX6 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Conjunctivochalasis (Eye disorders) | 0 | 1
Corneal epithelium defect (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 1
Limbal stem cell deficiency (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 2
Pinguecula (Eye disorders) | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Oral pain (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 8
Feeling cold (General disorders) | 0 | 3
Infusion site pain (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 3
Conjunctivitis (Infections and infestations) | 0 | 1
Dermatophytosis of nail (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CTA generally does not restrict an investigator's discussion of trial results after completion. Amgen has limited time to review material discussing trial results (up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control/approval of content. For multicenter studies, PI agrees not to publish results before first multi-center publication for at least 18 mo after study completion at all sites & all analyses of data resulting from Study.

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03343301/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03343301/SAP_001.pdf